CLINICAL TRIAL: NCT04590430
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose First-in-Human Study Investigating the Safety, Tolerability, and Pharmacokinetics of Intravenously Administered HFB30132A, a Monoclonal Antibody Directed Against SARS-CoV-2, in Healthy Adult Subjects
Brief Title: Study to Assess the Safety, Tolerability, and Pharmacokinetics of HFB30132A Against COVID-19 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HiFiBiO Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HFB30132A-101
Record Dates: First submitted 2020-10-08; First posted 2020-10-19 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Healthy
MeSH Terms: interventions — enuzovimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HFB30132A (Experimental): Participants will receive HFB30132A administered across 3 fixed-dose cohorts via intravenous infusions (to be administered sequentially)
  Interventions: Drug: HFB30132A
- Placebo (Placebo Comparator): Placebo will be administered to participants across three fixed-dose cohorts similar to the active treatment.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: HFB30132A — Participants randomized to HFB30132A will be administered dose 1 in cohort 1. Participants in Cohort 2 and 3 will receive HFB30132A doses 2 and 3, respectively.
  Arms: HFB30132A
Other: Placebo — Participants randomized to placebo will receive the same volume of solution as participants on active treatment.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the safety and tolerability of HFB30132A when it is given by intravenously to healthy participants. Blood tests will be done to check how much HFB30132A is in the bloodstream and how long the body takes to eliminate it. Participation may include up to ten visits to the study center.

DETAILED DESCRIPTION:
This is a Phase I, first time in human, randomized, double-blind, placebo-controlled, and dose escalation study in healthy volunteers.

The study will comprise of:

1. A Screening Period of up to 30 days (Day -30 through Day -1);
2. A Treatment Period during which participants will be resident at the Observation Unit from Day -1, 1 day before Investigational Medicinal Product (IMP) administration (on Day 1) until at least 24 hours after IMP administration, will be discharged on Day 2 after all safety and/or pharmacokinetic (PK) evaluations have been completed, and
3. A Follow up Period lasting 180 days after the IMP dose. The study will be conducted at a single study center in Cincinnati.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a healthy male or female subject, aged between 18 to 60 years (both inclusive). Health is defined as no clinically relevant abnormalities identified by Investigator's decision based on a detailed medical history, full physical examination, including blood pressure, heart rate, respiratory rate, and body temperature measurement, electrocardiogram (ECG) and clinical laboratory tests prior to the study drug administration.
* Subject is confirmed as negative by SARS-CoV-2 RT-PCR testing on screening and prior to admission to the unit.
* Subject voluntarily agrees to participate in this study and has given written informed consent prior to undergoing any of the screening procedures.
* Willing and able to comply with all scheduled visits, treatment plan, clinical laboratory tests, lifestyle guidelines, methods of contraception, including COVID-19 social distancing guidelines as described in Section 5.7.2 (under "Hygiene") from signing of informed consent through end of study on Day 180.
* Female subjects of childbearing potential must not be planning a pregnancy or be pregnant or lactating. All female subjects must have a negative result for the pregnancy tests performed at screening and admission.
* Female subjects of childbearing potential (including perimenopausal females who have had a menstrual period within 1 year prior to screening) must agree to use a reliable method of contraception until study completion and for at least 4 weeks following their final study visit on Day 180. Reliable contraception is defined as a method which results in a low failure rate, i.e., less than 1% per year when used consistently and correctly, such as hormonal contraception (oral, implant, injection, ring, or patch) and intrauterine contraceptive devices (IUDs) at least 3 months prior to Screening or a vasectomized partner. Note: Complete abstinence from sexual intercourse is acceptable.
* Female subject is of non-childbearing potential defined as surgically sterile (i.e. documented bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or at least 12 months postmenopausal (defined with no menses without an alternative medical cause and follicle stimulating hormone test in the post-menopausal range at the screening visit.
* Male subjects with partners of childbearing potential must have had surgical sterilization (vasectomy) at least 26 weeks prior to screening or use a male barrier method of contraception (i.e. male condom with spermicide) during any sexual intercourse, from Study Day -1 (beginning of confinement) until 3 months after the final Follow-up Visit on Day 270. Note: complete abstinence from sexual intercourse is acceptable.
* Male subjects must agree to abstain from sperm donation from initial study drug administration through 3 months after the last Follow-up Visit on Day 180.

Exclusion Criteria:

* History of any illness or history or presence of clinically significant pathology that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug(s) to the subject or collecting samples for analysis. This includes, but is not limited to, a history of relevant drug or food allergies; history of clinically significant cardiovascular, pulmonary, autoimmune, psychiatric or central nervous system disease, or of cancer with systemic spread in remission for less than 5 years.
* Use of any medications started within 14 days (or 5 half-lives, whichever is longer) prior to study drug administration including, prescription medications, nutritional supplements, and over-the-counter medications except for vitamin supplements, hormonal contraception, and recommended doses of acetaminophen, aspirin or ibuprofen
* Hospitalization for any reason within 60 days prior to the screening visit
* History of or positive human immunodeficiency virus (HIV) screen result, or positive blood test for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb). Subjects with positive hepatitis C virus (HCV) antibody at the screening visit are only eligible if they have previously completed treatment for HCV and have confirmatory negative test for HCV RNA.
* History of drug or alcohol abuse within 1 year prior to screening, or positive test for drugs of potential abuse at screening and admission, where alcohol abuse is defined as regular consumption exceeding 7 drinks/ week for women, and 14 drinks/ week for men.
* Participation (defined as receipt of dose of investigational agent) in any clinical research study evaluating another investigational drug or therapy within 30 days or at least 5 half-lives (whichever is longer), of the investigational drug prior to the screening visit
* Blood donation of approximately 1 pint (500 mL) within 60 days prior to dosing, or donation of more than 1 unit of plasma within 30 days prior to the start of study drug dosing
* Receipt of any transfused blood products within 60 days of the screening visit.
* Any history of receiving treatment or vaccination against SARS-CoV-2
* Febrile illness within 28 days prior to the first dose of study drug, or other signs or symptoms consistent with SARS-CoV-2 infection in the judgement of the Investigator in the 14 days prior to the first dose of study drug.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent serious adverse events (TESAEs) | From Day 1 to up to Day 30 of the last enrolled subject
  Number of participants experiencing TEAEs
Number of participants with treatment emergent adverse events (TEAE) of special interest | From Day 1 to up to Day 30 of the last enrolled subject
  Safety and tolerability will be evaluated in terms of number of participants with TEAEs of special interest (hypersensitivity / anaphylactic reaction / local tolerability)
Number of participants with treatment-emergent adverse events (TEAE) | From Day 1 to up to Day 30 of the last enrolled subject
  Safety and tolerability will be evaluated in terms of number of participants with TEAE
Maximum observed serum concentration (Cmax) | From Day 1 to up to Day 30 of the last enrolled subject
Minimum observed serum concentration (Cmin) | From Day 1 to up to Day 30 of the last enrolled subject
Time of maximum serum concentration (Tmax) | From Day 1 to up to Day 30 of the last enrolled subject
Area under the concentration vs. time curve (AUC0-last), AUC0-∞) | From Day 1 to up to Day 30 of the last enrolled subject
Terminal half-life (T1/2) | From Day 1 to up to Day 30 of the last enrolled subject
Systemic clearance (CL) | From Day 1 to up to Day 30 of the last enrolled subject
Steady-state volume of distribution (Vss) | From Day 1 to up to Day 30 of the last enrolled subject

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | From Day 1 to up to last follow-up day (Day 180)
  Safety and tolerability will be evaluated in terms of number of participants with TEAEs
Number of participants with treatment-emergent serious adverse events (TESAEs) | From Day 1 to up to last follow-up day (Day 180)
  Safety and tolerability will be evaluated in terms of number of participants with TESAEs
Maximum observed serum HFB30132A concentration (Cmax) in nasal and oral secretions | From Day 1 to up to last follow-up day (Day 180)
Minimum observed serum HFB30132A concentration (Cmin) in nasal and oral secretions | From Day 1 to up to last follow-up day (Day 180)
Time of maximum serum HFB30132A concentration (Tmax) in nasal and oral secretions | From Day 1 to up to last follow-up day (Day 180)
Area under the concentration vs. time curve (AUC0-last), AUC0-∞) in nasal and oral secretions | From Day 1 to up to last follow-up day (Day 180)
Terminal half-life (T1/2) of HFB30132A in nasal and oral secretions | From Day 1 to up to last follow-up day (Day 190)
Systemic clearance (CL) of HFB30132A in nasal and oral secretions | From Day 1 to up to last follow-up day (Day 180)
Steady-state volume of distribution (Vss) of HFB30132A in nasal and oral secretions | From Day 1 to up to last follow-up day (Day 180)
HFB30132A Anti-drug antibodies | From Day 1 to up to last follow-up day (Day 180)
  Presence or absence of antibodies against HFB30132A over time

CONTACTS AND LOCATIONS:
Overall Officials: Leela Vrishabhendra, MD, Principal Investigator — Medpace, Inc.
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen Y, Li S, Hedrich W, Wu X, Li S, Qiu C, Lin K, Bian X, He J, Zhou H, Adrian F, Schweizer L, Zhang J. Population pharmacokinetics and pharmacodynamics of HFB30132A, a monoclonal antibody against SARS-CoV-2, in healthy Chinese and US subjects. Int J Antimicrob Agents. 2025 Mar;65(3):107439. doi: 10.1016/j.ijantimicag.2024.107439. Epub 2025 Jan 9. PMID 39793935
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343